CLINICAL TRIAL: NCT04519853
Title: A Pilot Study to Test the Safety and Tolerability of a Low Glycemic Load Dietary Intervention in Adults With Cystic Fibrosis
Brief Title: A Pilot Study of a Low Glycemic Load Diet in Adults With Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Melissa Putman, Assistant Professor of Pediatrics, Attending in Endocrinology, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P00034904
Record Dates: First submitted 2020-07-07; First posted 2020-08-20 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Cystic Fibrosis; Cystic Fibrosis-related Diabetes; Cystic Fibrosis With Intestinal Manifestations
Keywords: Cystic Fibrosis Related Diabetes; Low Glycemic Load; Continuous Glucose Monitoring
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Intervention Model Description: Single dietary treatment arm with run-in period as a control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low Glycemic Load Diet (Experimental): Feeding study with dietary composition (approximately) 50% fat, 30% carbohydrate, 20% protein.
  Interventions: Behavioral: Low Glycemic Load Diet

INTERVENTIONS:
Behavioral: Low Glycemic Load Diet — Food delivery service will provide a low glycemic load diet for 8 weeks

SUMMARY:
This pilot study will evaluate the safety and tolerability of a low glycemic load dietary intervention in adult patients with cystic fibrosis (CF) in a rigorous feeding study. Specific emphasis will be placed on changes in weight, body composition, and glycemic measures obtained via continuous glucose monitor (CGM) usage.

DETAILED DESCRIPTION:
Non-pulmonary complications of cystic fibrosis (CF) are becoming increasingly prevalent with the changing landscape of CF care. CF related diabetes mellitus (CFRD) and CF related gastrointestinal (GI) complications have significant effects on morbidity and mortality. Treatment options are limited to insulin therapy for CFRD and symptom control for most GI complications.

BMI is a well-established marker of morbidity and mortality in patients with CF. Many patients consume a high carbohydrate intake to meet their increase caloric needs, potentially leading to complications including post-prandial hyperglycemia, increased inflammation, and abnormal GI motility. Dietary recommendations for children and adults with CF are limited and based entirely on consensus and expert opinion. As patients with CF live longer with highly effective modulator therapy, it is important to understand the effects of dietary composition on short and long-term endocrine, GI, and pulmonary outcomes.

The investigators will conduct a prospective, open-label pilot study in adults with CF and impaired glucose tolerance or indeterminate glycemia to establish the safety and tolerability of a low glycemic load (LGL) diet. Subjects will initially follow their standard diet for a 2-week run-in period, then transition to a LGL diet provided by a food delivery service for the remaining 8 weeks. The investigators will also investigate potential short-term outcomes of dietary carbohydrate manipulation, including glycemic variability measured by continuous glucose monitor (CGM), body composition via DXA, GI symptoms, and quality of life measures.

The investigators hypothesize that a diet lower in carbohydrate content will be safe, tolerable, and associated with weight maintenance or gain, and that a LGL diet will result in decreased glycemic variability via CGM, improved GI symptoms, increased lean to fat mass ratio, and improved quality of life measures over an 8-week period.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of CF
2. Diagnosis of pancreatic insufficiency, requiring pancreatic enzyme replacement
3. Oral glucose tolerance test within the past three years showing impaired glucose tolerance (2-hour glucose ≥140 mg/dL) or indeterminate glycemia (1-hour glucose ≥200), HbA1c 5.7-6.4% in the past one year, and/or or documented random glucose ≥200 in the past one year
4. BMI 21-25 kg/m2
5. 18 years and above

Exclusion Criteria:

1. Current use of insulin
2. Most recent HbA1c ≥6.5%
3. History of solid organ transplant or currently listed for solid organ transplant
4. FEV1 <50% predicted on most recent pulmonary function testing
5. Currently receiving enteral nutrition support
6. Current or anticipated pregnancy in the next 1 year
7. Hospitalization for CF exacerbation within 1 month of enrollment
8. Started or stopped treatment with Trikafta or other CFTR modulator within 3 months of enrollment
9. Currently adhering to a low glycemic index or other carbohydrate restricted diet

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Change in weight from baseline and 10 weeks | Baseline and 10 weeks
  Anthropometric measure
Change in percent time <54 mg/dL | Baseline and 10 weeks
  Continuous glucose monitoring
Patient reported tolerability of dietary intervention, Likert scale | Single measurement at 10 weeks after diet completion
  Single Likert scale question of overall diet tolerability, ranging from 1 (intolerable) to 10 (completely tolerable)

SECONDARY OUTCOMES:
Change in percent time >140 mg/dL | Baseline to 10 weeks
  Continuous glucose monitoring
Change in CGM average glucose | Baseline to 10 weeks
  Continuous glucose monitoring
Change in CGM glucose management indicator (GMI) | Baseline to 10 weeks
  Continuous glucose monitoring
Change in CGM standard deviation (SD) | Baseline to 10 weeks
  Continuous glucose monitoring
Change in CGM coefficient of variation (CV) | Baseline to 10 weeks
  Continuous glucose monitoring
Change in percent time less than 50 mg/dL on CGM | Baseline to 10 weeks
  Continuous glucose monitoring
Change in percent time less than 70 mg/dL on CGM | Baseline to 10 weeks
  Continuous glucose monitoring
Change in percent time 70-180 mg/dL on CGM | Baseline to 10 weeks
  Continuous glucose monitoring
Change in percent time greater than 180 mg/dL on CGM | Baseline to 10 weeks
  Continuous glucose monitoring
Change in percent time greater than >250 mg/dL on CGM | Baseline to 10 weeks
  Continuous glucose monitoring
Number of episodes of symptomatic hypoglycemia | Baseline and 10 weeks
  Survey
Change in lean and fat mass | Baseline and 10 weeks
  DXA body composition measures
Change in Patient Assessment of Constipation (PAC) questionnaire score | Baseline and 10 weeks
  Likert scale questionnaire with 12 items, each item scored 0-4, total score ranging from 0-48 with higher scores related to worse outcomes
Change in Patient Assessment of Gastrointestinal Symptom (PAGI-SYM) questionnaire score | Baseline and 10 weeks
  Likert scale questionnaire with 20 items, each item scored 0-5, total score ranging from 0-100 with higher scores related to worse outcomes
Change in Modified Activity Questionnaire (MAQ) score | Baseline and 10 weeks
  Questionnaire, units of total hours of exercise over past 12 months, no min or max scores, higher value related to better outcome
Change in Cystic Fibrosis Questionnaire Revised (CFQ-R) score | Baseline and 10 weeks
  Likert scale questionnaire, 50 items, each scored 0-4, total score ranging from 0-100 with higher value reflecting better outcome
Change in erythrocyte sedimentation rate (ESR) | Baseline and 10 weeks
  Laboratory test, measured in mm/hr
Change in c-reactive protein (CRP) | Baseline and 10 weeks
  Laboratory test, measured in mg/L
Change in intestinal fatty acid binding protein (I-FABP) | Baseline and 10 weeks
  Laboratory test, measured in ng/mL

CONTACTS AND LOCATIONS:
Overall Officials: Melissa S Putman, MD,MS, Principal Investigator — Boston Children's Hospital; Massachusetts General Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD data with other researchers.

REFERENCES:
- [Background] Moran A, Brunzell C, Cohen RC, Katz M, Marshall BC, Onady G, Robinson KA, Sabadosa KA, Stecenko A, Slovis B; CFRD Guidelines Committee. Clinical care guidelines for cystic fibrosis-related diabetes: a position statement of the American Diabetes Association and a clinical practice guideline of the Cystic Fibrosis Foundation, endorsed by the Pediatric Endocrine Society. Diabetes Care. 2010 Dec;33(12):2697-708. doi: 10.2337/dc10-1768. No abstract available. PMID 21115772
- [Background] Gabel ME, Galante GJ, Freedman SD. Gastrointestinal and Hepatobiliary Disease in Cystic Fibrosis. Semin Respir Crit Care Med. 2019 Dec;40(6):825-841. doi: 10.1055/s-0039-1697591. Epub 2019 Oct 28. PMID 31659728
- [Background] Prentice BJ, Ooi CY, Strachan RE, Hameed S, Ebrahimkhani S, Waters SA, Verge CF, Widger J. Early glucose abnormalities are associated with pulmonary inflammation in young children with cystic fibrosis. J Cyst Fibros. 2019 Nov;18(6):869-873. doi: 10.1016/j.jcf.2019.03.010. Epub 2019 Apr 26. PMID 31036487
- [Background] Brennan AL, Gyi KM, Wood DM, Johnson J, Holliman R, Baines DL, Philips BJ, Geddes DM, Hodson ME, Baker EH. Airway glucose concentrations and effect on growth of respiratory pathogens in cystic fibrosis. J Cyst Fibros. 2007 Apr;6(2):101-9. doi: 10.1016/j.jcf.2006.03.009. Epub 2006 Jul 17. PMID 16844431
- [Background] Balzer BW, Graham CL, Craig ME, Selvadurai H, Donaghue KC, Brand-Miller JC, Steinbeck KS. Low glycaemic index dietary interventions in youth with cystic fibrosis: a systematic review and discussion of the clinical implications. Nutrients. 2012 Apr;4(4):286-96. doi: 10.3390/nu4040286. Epub 2012 Apr 18. PMID 22606371